CLINICAL TRIAL: NCT02546661
Title: An Open-Label, Randomised, Multi-Drug, Biomarker-Directed, Multi-Centre, Multi-arm Phase 1b Study in Patients With Muscle Invasive Bladder Cancer (MIBC) Who Have Progressed on Prior Treatment (BISCAY).
Brief Title: Open-Label, Randomised, Multi-Drug, Biomarker-Directed, Phase 1b Study in Pts w/ Muscle Invasive Bladder Cancer
Acronym: BISCAY
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2615C00001; GU 118 (Other: Sarah Cannon Development Innovations, LLC); BISCAY (Other: Sponsor); 2015-002228-25 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-11 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Durvalumab; Olaparib; Vistusertib; Selumetinib; Muscle invasive bladder cancer; MIBC; BISCAY; MEDI4736; AZD4547; AZD2281; AZD1775; AZD2014; AZD9150; AZD6244
MeSH Terms: interventions — AZD4547; durvalumab; olaparib; adavosertib; vistusertib; danvatirsen; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Module A: AZD4547 Monotherapy (Experimental): AZD4547 will be given orally twice daily until disease progression.
  Patients who receive AZD4547 as monotherapy will have the option to cross over to durvalumab as monotherapy at the point of objective progression, as long as the following criteria are met:
  * The investigator believes it is in the patient's interest to receive durvalumab;
  * The patient consents to the continued treatment;
  * It is clinically appropriate for the patient to continue on durvalumab treatment;
  * The patient satisfies the key eligibility criteria for receiving durvalumab treatment.
  Interventions: Drug: AZD4547
- Module A: MEDI4736 (durvalumab) + AZD4547 (Experimental): AZD4547 will be given orally twice daily until disease progression. Patients will also receive MEDI 4736 (durvalumab) by IV infusion once every 4 weeks.
  Interventions: Drug: AZD4547; Drug: MEDI4736
- Module B: MEDI4736 (durvalumab) + Olaparib (Experimental): MEDI4736 (durvalumab) will be given by IV infusion once every 4 weeks. Olaparib will be given orally twice daily.
  Interventions: Drug: MEDI4736; Drug: Olaparib
- Module C: MEDI4736 (durvaluamb) + AZD1775 (Experimental): MEDI4736 (durvalumab) will be given by IV infusion once every 4 weeks. AZD1775 will be given orally in approximate 12 hour intervals over 3 days (6 doses) on Days 1-3, 8-10, and 15-17 of 28 day cycles.
  Interventions: Drug: MEDI4736; Drug: AZD1775
- Module D: MEDI4736 (durvalumab) monotherapy (Experimental): MEDI 4736 (durvalumab) will be given by IV infusion once every 4 weeks.
  Interventions: Drug: MEDI4736
- Module E: MEDI4736 (durvalumab) + Vistusertib (Experimental): MEDI4736 (durvalumab) will be given by IV infusion once every 4 weeks. Vistusertib will be given orally twice per day on an intermittent schedule (2 days on, 5 days off).
  Interventions: Drug: MEDI4736; Drug: Vistusertib
- Module F: MEDI4736 (durvaluamb) + AZD9150 (Experimental): AZD9150 will be given as monotherapy on Days -7, -5, and -3 of a one week lead-in period. Combination dosing with IV AZD9150 followed by IV MEDI4736 (durvalumab) begins on Day 1 of each 28 day cycle. Thereafter AZD9150 is given weekly and MEDI4736 is given once every 4 weeks.
  Interventions: Drug: MEDI4736; Drug: AZD9150
- Module G: MEDI4736 + Selumetinib (Experimental)
  Interventions: Drug: MEDI4736; Drug: Selumetinib

INTERVENTIONS:
Drug: AZD4547 — AZD4547 Monotherapy vs. MEDI4736 (durvalumab) + AZD4547 1:1 Randomization.
  Arms: Module A: AZD4547 Monotherapy; Module A: MEDI4736 (durvalumab) + AZD4547
Drug: MEDI4736 — MEDI4736
  Other Names: Durvalumab
  Arms: Module A: MEDI4736 (durvalumab) + AZD4547; Module B: MEDI4736 (durvalumab) + Olaparib; Module C: MEDI4736 (durvaluamb) + AZD1775; Module D: MEDI4736 (durvalumab) monotherapy; Module E: MEDI4736 (durvalumab) + Vistusertib; Module F: MEDI4736 (durvaluamb) + AZD9150; Module G: MEDI4736 + Selumetinib
Drug: Olaparib — MEDI4736 (durvalumab) + Olaparib
  Other Names: Lynparza
  Arms: Module B: MEDI4736 (durvalumab) + Olaparib
Drug: AZD1775 — MEDI4736 (durvalumab) + AZD1775
  Arms: Module C: MEDI4736 (durvaluamb) + AZD1775
Drug: Vistusertib — MEDI4736 (durvalumab) + Vistusertib
  Arms: Module E: MEDI4736 (durvalumab) + Vistusertib
Drug: AZD9150 — MEDI4736 (durvalumab) + AZD9150
  Arms: Module F: MEDI4736 (durvaluamb) + AZD9150
Drug: Selumetinib — MEDI4736 (durvalumab) + Selumetinib
  Arms: Module G: MEDI4736 + Selumetinib

SUMMARY:
This is an open label, multi-drug, biomarker-directed, multi-centre, multi-arm, Phase 1b study in patients with muscle invasive bladder cancer (MIBC) (urothelial) who have progressed on prior treatment. This study is modular in design, allowing evaluation of the safety, tolerability, pharmacokinetics and anti-tumour activity of multiple agents as monotherapy and as combinations of different novel anti-cancer agents.

The study will consist of a number of study modules (sub-studies), each evaluating the safety and tolerability of a specific agent or combination.

DETAILED DESCRIPTION:
This is an open label, multi-drug, biomarker-directed, multi-centre, multi-arm, Phase 1b study in patients with muscle invasive bladder cancer (MIBC) (urothelial) who have progressed on prior treatment. This study is modular in design, allowing evaluation of the safety, tolerability, pharmacokinetics and anti-tumour activity of multiple agents as monotherapy and as combinations of different novel anti-cancer agents.

The study will consist of a number of study modules (sub-studies), each evaluating the safety and tolerability of a specific agent or combination in patients whose tumours express specific genomic alterations relevant to the molecules under investigation and whose disease has progressed following prior therapy. The allocation of patients to specific modules will depend on the specific eligible genomic alterations identified in their tumours.

Each module will determine the appropriate combination dose for further clinical evaluation based on safety, tolerability and efficacy profile. A maximum tolerated dose will be defined and each arm expanded appropriately to explore further the safety, tolerability, pharmacokinetics and biological activity at the selected combination doses.

Module A includes an AZD4547 monotherapy arm and a MEDI4736 (durvalumab) + AZD4547 combination therapy arm and will investigate the safety and tolerability of MEDI4736 given intravenously, in combination with AZD4547 given orally to selected patients with MIBC with tumours that have fibroblast growth factor receptor mutations or fibroblast growth factor receptor fusions.

Module B will investigate the safety and tolerability of MEDI4736 given intravenously in combination with olaparib (AZD2281, Lynparza) given orally to selected patients with MIBC whose tumors have mutations in a homologous recombination repair gene panel and whose disease had progressed following prior therapy.

Module C will investigate the safety and tolerability of MEDI4736 given intravenously, in combination with AZD1775 given orally to selected patients with MIBC whose tumours have mutations in genes involved in cell cycle regulation (e.g., loss of either retinoblastoma 1 or cyclin-dependent kinase inhibitor 2A or amplification of cyclin E1 or MYC family genes).

Module D will investigate the safety and tolerability of MEDI4736 given intravenously as monotherapy to patients with MIBC who do not qualify for Modules A, B or C.

Module E will investigate the safety and tolerability of MEDI4736 given intravenously, in combination with vistusertib (AZD2014) given orally to patients with MIBC whose tumours do not show genomic alterations that would be eligible for other study modules. Patients whose MIBC tumours harbour the following genomic alterations that have potential to respond to a mammalian target of rapamycin (mTOR) inhibitor will also be included in Module E: RICTOR amplification, or TSC1/1 mutations.

Module F will investigate the safety and tolerability of MEDI4736 given intravenously in combination with AZD9150 given intravenously to patients with MIBC whose tumours do not show genomic alterations that would be eligible for other modules.

Module G will investigate the safety and tolerability of MEDI4736 given intravenously in combination with selumetinib (AZD6244) given orally to patients with MIBC. Patients in this module will not be selected for any specific tumour genomic alteration.

ELIGIBILITY:
Inclusion Criteria for all Modules:

1. Metastatic MIBC
2. 2nd/3rd line
3. Failed adjuvant/neo-adjuvant chemotherapy <1 yr
4. 1 lesion ≥10 mm at baseline in the longest diameter suitable for accurate repeated measurement
5. WHO perf. status 0-1

For Module A:

1. M/F ≥25
2. Confirmation of FGFR3 mutation or FGFR fusion

For Module B:

1. Hgb ≥10 g/dL
2. Deleterious mutation, deletion or truncation in any HRR genes

For Module C:

1. Tumour harbours a deletion or inactivating mutation of the CDKN2A or RB1 genes and/or amplification of CCNE1, MYC, MYCL or MYCN genes

For Module E:

1. Contraception must be sustained throughout treatment with vistusertib and 16 wks after last dose

For Module F:

1. Adequate organ and marrow function, defined as Leukocytes ≥3.0x10(exp9)/L; ANC ≥1.5x10(exp9)/L; platelets ≥100x10(exp9)/L
2. Contraceptive measures must be sustained throughout treatment with AZD9150 and for 180 days after the last dose.

Exclusion Criteria for all Modules:

1. Immunotherapy, chemotherapy, anticancer agents, radiotherapy <4 weeks, or radiotherapy for palliation <2 weeks, any study drugs <30 days.
2. Major surgery <4 weeks
3. Unresolved toxicities from prior therapy
4. Concurrent chemotherapy, immunotherapy, biologic or hormonal therapy
5. Immunosuppressive drugs <28 days
6. Any of the following: Autoimmune disease ≤2 yr; IBD; primary immunodeficiency; organ transplant requiring immunosuppressives
7. Spinal cord compression or brain metastases, treated and stable & not requiring steroids for at least 4 weeks
8. Severe or uncontrolled systemic disease
9. Any of the following: Mean QTc ≥470 ms; abnormalities in resting ECG; factors that increase the risk of QTc prolongation or arrhythmia; uncontrolled hyper/hypotension; LVEF <55%; atrial fibrillation; NYHA Grade II-IV; severe valvular disease; uncontrolled angina; stroke/TIA <6 months; acute coronary syndrome <6 months
10. Any of the following laboratory values: ANC <1.5x10(exp9)/L; Platelets <100x10(exp9)/L; Hgb <9.0 g/dL; ALT >2.5xULN or >5xULN with liver mets; Total bilirubin >1.5 times ULN or with Gilbert's disease ≥2×ULN; Creatinine >1.5xULN concurrent with creatinine clearance <50 mL/min; Corrected Ca >ULN, PO4 >ULN
11. Active infection including tuberculosis, hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus. Patients with a past or resolved HBV infection are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Live attenuated vaccination <30 days

For Module A:

1. Prior exposure to: Nitrosourea or mitomycin C <6 weeks; any agent with FGFR inhibition as its primary pharmacology; AZD4547; potent inhibitors/inducers of CYP3A4, inhibitors of CYP2D6 or substrates of CYP3A4 <2 wks
2. Ophthalmological criteria: RPED; laser treatment or intraocular injection for macular degeneration; age-related macular degeneration; retinal vein occlusion; retinal degenerative disease; other clinically relevant chorioretinal defect
3. Refractory nausea/vomiting, chronic GI diseases, or previous bowel resection

For Module B:

1. Transfusion <120 days
2. Concurrent medications that are strong inhibitors of cytochrome P450 (CYP) 3A (CYP3A) or strong inducers of CYP3A4.
3. Previous treatment with PARP inhibitor, including olaparib
4. Patients with history of MDS or AML

For Module C:

1. Prior exposure to any of the following: Nitrosourea or mitomycin C <6 wks; any agent with Wee1 inhibition as its primary pharmacology; prior treatment with AZD1775
2. Any drugs or products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with narrow therapeutic index, or moderate to strong inhibitors/inducers of CYP3A4
3. Herbal preparations
4. Refractory nausea and vomiting or chronic GI diseases
5. Cardiac disease <6 months

For Module E:

1. Minor surgery <14 days of first dose
2. Exposure to specific substrates of OATP1B1, OATP1B3, MATE1 and MATE2K <5x half-life before treatment. Exposure to strong/moderate inhibitors/inducers of CYP3A4/5, Pgp (MDR1) and BRCP if taken within washout periods before the first dose
3. Haemopoietic growth factors (filgrastim, sargramostim, GM-CSF) <14 days prior to treatment
4. Other mTOR inhibitors
5. Renal disease or renal tubular acidosis
6. Uncontrolled Type 1 or 2 diabetes

For Module F:

1. AST ≤ 2.5xULN or ≤5xULN with liver metastases

For Module G:

1. Have had prior treatment with a MEK, Ras or Raf inhibitor.
2. Any of the following ophthalmic criteria: Current or past history of central serous retinopathy, detachment of retinal pigmented epithelium, or retinal vein occlusion; intraocular pressure (IOP) >21 mmHg; uncontrolled glaucoma (irrespective of IOP)
3. Baseline left ventricular ejection fraction (LVEF) <55% measured by echocardiogram (ECHO) or, if allowed, a multigated acquisition (MUGA) scan. Appropriate correction to be used if a MUGA is performed.
4. Previous moderate or severe impairment of LVEF (<45% on echocardiography or equivalent on MUGA) even if full recovery has occurred.
5. Male or female patients with reproductive potential and, as judged by the investigator, are not employing an effective method of birth control and female patients who are breastfeeding.
6. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
7. Receiving or have received systemic therapy with nitrosoureas, mitomycin or suramin within 6 weeks prior to starting study treatment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Module A: The frequency and nature of adverse events related to AZD4547 monotherapy. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of AZD4547 monotherapy given orally to selected patients with MIBC who have progressed following prior therapy.
Module A: The frequency and nature of adverse events related to the combination of intravenous MEDI4736 (durvalumab) and oral AZD4547. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI4736 (durvalumab) given intravenously in combination with AZD4547 given orally to selected patients with MIBC who have progressed following prior therapy.
Module B: The frequency and nature of adverse events related to the combination of intravenous MEDI4736 (durvalumab) and oral olaparib. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI4736 (durvalumab) given intravenously in combination with olaparib given orally to selected patients with MIBC who have progressed following prior therapy.
Module C: The frequency and nature of adverse events related to intravenous MEDI4736 (durvalumab) when given in combination with oral AZD1775. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI4736 (durvalumab) given intravenously in combination with AZD1775 given orally to selected patients with MIBC who have progressed following prior therapy.
Module D: The frequency and nature of adverse events related to intravenous MEDI4736 (durvalumab) monotherapy. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI4736 (durvalumab) monotherapy given intravenously to selected patients with MIBC who have progressed following prior therapy.
Module E: The frequency and nature of adverse events related to intravenous MEDI4736 (durvalumab) when given in combination with oral vistusertib. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI 4736 (durvalumab) given intravenously in combination with vistusertib given orally to selected patients with MIBC who have progressed following prior therapy.
Module F: The frequency and nature of adverse events related to the combination of intravenous MEDI4736 (durvalumab) and intravenous AZD9150. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of intravenous MEDI4736 (durvalumab) in combination with intravenous AZD9150 in selected patients with MIBC who have progressed following prior therapy.
Module G: The frequency and nature of adverse events related to intravenous MEDI4736 (durvalumab) when given in combination with oral selumetinib. | Adverse events will be assessed at each clinic visit, and at study discontinuation and 90 days after the end of treatment. Clinic visits are generally scheduled weekly.
  The frequency and nature of adverse events will be assessed in order to determine the safety and tolerability of MEDI 4736 (durvalumab) given intravenously in combination with selumetinib given orally to selected patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in clinical chemistry parameters. | Days 1, 8, 15, and 22 of Cycle 1, Days 1, 15, and 22 of Cycles 2 and 3 and every 4 weeks thereafter, and at discontinuation.
  Changes from baseline in clinical chemistry parameters will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in haematology parameters. | Days 1, 8, 15, and 22 of Cycle 1, Days 1, 15, and 22 of Cycles 2 and 3 and every 4 weeks thereafter, and at discontinuation.
  Changes from baseline in haemotology parameters will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in urinalysis results. | Days 1, 8, 15, and 22 of Cycle 1, Days 1, 15, and 22 of Cycles 2 and 3 and every 4 weeks thereafter, and at discontinuation.
  Changes from baseline in urinalysis findings will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in vital signs. | Day 1 of Cycles 1, 2, 3, and 4 and every 4 weeks therafter, and at discontinuation.
  Changes from baseline in vital signs will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in physical examination findings. | Day 1 of Cycles 1, 2, 3, and 4 and every 4 weeks therafter, and at discontinuation.
  Changes from baseline in physical examination findings will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in ECG findings. | ECGs will be collected at screening, Day 1, Cycle 1and then Day 1 of each cycle from Cycle 2 onwards.
  Changes from baseline in ECG findings will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in ejection fraction determined by assessing ECHO/MUGA scans. | Ejection fraction will be measured at screening, on Day 1, Cycle 1, and every 12 weeks thereafter (relative to the first dose of study drug) up to Cycle 7, and then every 16 weeks thereafter.
  Changes from baseline in ejection fraction determined by assessing ECHO/MUGA scans will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in coagulation parameters | Coagulation parameters will be measured at screening, on Day 1, Cycle 1, and every 12 weeks thereafter (relative to the first dose of study drug) up to Cycle 7, and then every 16 weeks thereafter.
  Changes from baseline in coagulation parameters will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.
All Modules: Change from baseline in lipid profile | Lipid profile will be measured at screening, on Day 1, Cycle 1, and every 12 weeks thereafter (relative to the first dose of study drug) up to Cycle 7, and then every 16 weeks thereafter.
  Changes from baseline in lipid profile will be assessed in order to determine the safety and tolerability of the drug regimen chosen in the sub study module for patients with MIBC who have progressed following prior therapy.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 16 weeks and 52 weeks
  The percentage of patients who have a confirmed visit response of Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST 1.1.
  Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be included in the assessment of ORR.
Disease control rate (DCR) | 16 weeks and 52 weeks
  Percentage of patients who have a confirmed visit response of CR or PR or stable disease (SD) ≥16 weeks as assessed by the investigator as per RECIST 1.1
Progression free survival (PFS) | up to 12 months
  The time from randomization until the date of objective disease progression or death (from any cause in the absence of progression) regardless of whether the patient withdraws from assigned therapy or receives another anticancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.
Duration of response (DoR) | up to 12 months
  Duration of response is defined as the elapsed time from the date of first documented response (CR/PR) as per RECIST Version 1.1 as assessed by the investigator until the date of documented progression or death in the absence of disease progression. The time of the initial response is defined as the latest of the dates contributing towards the first visit response of PR or CR.
Overall survival (OS) rate at 1 year | 1 year
  Defined as the proportion of patients surviving after 1 year from the start of treatment.
Plasma concentration of AZD4547 (Module A) | Blood samples will be taken pre-dose on Days 1 and 8 of Cycle 1; pre-dose and 2, 3, 4 and 6 hours post-dose on Day 1 of Cycle 2; and pre-dose and 2 to 4 hours post-dose on Day 1 of Cycle 3.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of MEDI4736 (durvalumab) (Module A) | Blood samples will be taken pre-dose and end of infusion for Day 1 of Cycles 1 to 7 and for the post-Cycle 7 8-weekly assessments, and pre-dose for Day 8 of Cycle 1.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of olaparib (Module B) | Blood samples will be taken on Day 3 of Cycles 1 and pre-dose and 4 hr post-dose. Serial samples on Day 3 of Cycle 3, pre-dose, 1, 2, 4, 6, 8, and 10 hr post-dose.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of AZD1775 (Module C) | Blood samples will be taken on Day 8 at steady state at the following time points: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hr post-dose.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of MEDI4736 (durvalumab) (Module C) | Blood samples will be taken on Days 1 and 8 of Cycle 1 pre-dose and at the end of infusion (1 hour). Samples will also be collected on Day 1 of Cycles 2 to 7 pre-dose and at the end of infusion.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of MEDI4736 (durvalumab) (Module D) | Blood samples will be taken on Days 1 and 8 of Cycle 1
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of vistusertib (Module E) | Blood samples will be collected pre-dose, and 2 and 4 hr post-dose on Day 1 of Cycle 1; and pre-dose and 2 to 6 hr post-dose (matched to biopsy) on Day 2 of Cycle 2.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of Medi4736 (durvalumab) (Module E). | Blood samples will be taken pre-dose and end of infusion for Day 1 of Cycles 1 to 7 and every 8 weeks thereafter and pre-dose for Day 8 of Cycle 1.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of AZD9150 (Module F) | Blood samples will be taken pre-dose of Days -7, -5, and -3 of the lead-in portion and thereafter prior to dosing and at the ned of infusion on Day 1 of Cycles 1, 2, 3, 4, 6, and 8 (approximately 8 months).
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
Plasma concentration of MEDI4736 (durvalumab) (Module F). | Blood samples will be taken pre-dose and end of infusion for Day 1 of Cycles 1 to 7 and every 8 weeks thereafter and pre-dose for Day 8 of Cycle 1.
  The timing of the PK samples may be adjusted during the study, dependent on emerging data, in order to ensure appropriate characterisation of the plasma concentration-time profiles.
The presence of Anti-Drug Antibodies (ADA) and ADA neutralising antibodies to MEDI4736 will be assessed in patients receiving MEDI4736 in any sub-study module. | Blood samples will be collected prior to MEDI4736 dosing on Day 1 of Cycles 1, 2 and 4 and every 12 weeks thereafter (up to 12 months).
  The formation of anti-drug antibodies and neutralizing antibodies will be assessed by validated methods.

OTHER OUTCOMES:
Mutation status of cancer associated genes in circulating tumour DNA (ctDNA). | Blood samples for assessment of ctDNA will be collected at screening, on Day 1 of Cycles 1, 2, 3, and 4 (up to 91 days) and at disease progression.
  Plasma and serum samples will be collected and assessed for circulating tumour DNA to explore the mutation status of cancer associated genes.
Biomarker Analysis of Blood and Tissue | Up to 12 months
  Biomarker analysis of blood and tissue to assess exploratory markers, which may include but is not limited to:
  * immune cell gene expression profiles and cytokine profiles within the peripheral and tumoural compartments,
  * the presence of IFN-γ, tumour necrosis factor-α, IL-2, IL-6, IL-10, IL-8, and IL-12 as well as antibodies against tumour, self, or viral antigens,
  * expression of PD-L1,
  * CD8 and the number and phenotype of immune cells such as T-cells.
  Markers relevant to the targeted therapy, for example FGFR and ligand expression and PD markers, for example pErk, pS6 and γH2AX will also be measured in tumour paired biopsy samples.
  Biomarker assessments that may have the potential to identify patients likely to respond to treatment with the agents studied in this modular protocol will be investigated to determine a patient's biomarker status and for possible correlation with efficacy endpoints.
Correlation of biomarkers to response and/or development of cancer | Throught out study (up to 18 months)
  To explore potential biomarkers in residual biological samples (e.g., tumour, plasma and/or serum) which may influence development of cancer (and associated clinical characteristics) and/or response.
Estimate overall survival (OS) | Up to 18 months
  To estimate the overall survival for patients have been pre-screened but do not enter the main part of the study.
Objective Response Rate (ORR) (by modified RECIST 1.1) | 16 weeks and 52 weeks
  The percentage of patients who have a confirmed response of CR or PR as assessed by the investigator using a modified RECIST 1.1. Modified RECIST 1.1 will be used for patients receiving MEDI4736 because of response may occur after progression has been initially determined. Patients receiving MEDI4736 may continue to receive treatment and be followed after an initial assessment of progression until subsequent confirmation. Confirmed progression is defined as ≥20% increase in sum of diameters of target lesions compared to the nadir at 2 consecutive visits; and/or significant progression (worsening) of non-target lesions (NTLs) or new lesions (NLs) at the confirmatory scan; and/or new unequivocal lesions at the confirmatory scan. If progression is not confirmed then the visit response is assessed as SD/PR or CR and the patient should continue scheduled scans. If progression is confirmed the visit response should be assessed as progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, MBBS, MRCP, MD, Principal Investigator — Barts Cancer Center, Barts and The London School of Medicine and Denistry; Hendrik-Tobias Arkenau, MD, PhD, Principal Investigator — Sarah Cannon Research Institute, UK
Locations (23):
- United States (6):
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Nashville, Tennessee
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (6):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Spain (3):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Powles T, Carroll D, Chowdhury S, Gravis G, Joly F, Carles J, Flechon A, Maroto P, Petrylak D, Rolland F, Cook N, Balar AV, Sridhar SS, Galsky MD, Grivas P, Ravaud A, Jones R, Cosaert J, Hodgson D, Kozarewa I, Mather R, McEwen R, Mercier F, Landers D. An adaptive, biomarker-directed platform study of durvalumab in combination with targeted therapies in advanced urothelial cancer. Nat Med. 2021 May;27(5):793-801. doi: 10.1038/s41591-021-01317-6. Epub 2021 May 3. PMID 33941921
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306
- See also: Clinical Study Protocol Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2615C00001&attachmentIdentifier=d31a0b6e-ec7a-461e-ab7d-2ec947a6da7c&fileName=CSP_Redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2615C00001&attachmentIdentifier=0d115291-20a8-4aa6-a33a-41e298985bf5&fileName=SAP_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2615C00001&attachmentIdentifier=b753b1dd-5e40-4eb0-bec7-141b1c2e1211&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: An adaptive, biomarker-directed platform study of durvalumab in combination with targeted therapies in advanced urothelial cancer — https://www.nature.com/articles/s41591-021-01317-6